CLINICAL TRIAL: NCT01387867
Title: Effects of Strength Training and Nordic Walking in Patients With Osteoarthritis of the Hip
Brief Title: Exercise in Patients With Osteoarthritis of the Hip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Nina Beyer, Assoc. Prof., Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOA-ISMC
Record Dates: First submitted 2011-06-29; First posted 2011-07-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2013-07

CONDITIONS: Hip Osteoarthritis
Keywords: Exercise; Hip osteoarthritis; Randomized controlled trial
MeSH Terms: conditions — Osteoarthritis, Hip; Motor Activity | interventions — Resistance Training; Nordic Walking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Strength training (Experimental): Strength training three times weekly, i.e.supervised strength training twice weekly and un-supervised strength training once weekly for 4 months.
  Interventions: Procedure: Strength training
- Nordic Walking (Experimental): Nordic walking three times weekly, i.e.Nordic walking twice weekly and un-supervised Nordic walking once weekly for 4 months.
  Interventions: Procedure: Nordic Walking
- Unsupervised home based exercise (Active Comparator): The home based unsupervised exercise comprised exercises recommended by the Danish Arthritis Association.
  Interventions: Procedure: Unsupervised home based exercise

INTERVENTIONS:
Procedure: Strength training — Supervised strength training in groups 2 x 1 hour weekly and un-supervised strength training 1 hour weekly for 4 months
  Arms: Strength training
Procedure: Nordic Walking — Supervised Nordic Walking in groups 2 x 1 hour weekly and un-supervised Nordic Walking 1 hour weekly for 4 months
  Arms: Nordic Walking
Procedure: Unsupervised home based exercise — Unsupervised home based exercise as recommended by the Danish Arthritis Association 1 hour 3 x weekly for 4 months
  Arms: Unsupervised home based exercise

SUMMARY:
According to Danish and international guidelines the recommended first-line of management for people with osteoarthritis consist of exercise, education, analgesic medication, and, if necessary, weight reduction. It is well documented that exercise has a positive effect on pain and physical function in patients with knee OA, but the effect of exercise on hip OA is sparsely investigated.

Aim of the study: To investigate the effects of 1) strength training, and 2) Nordic Walking, and 3) unsupervised home based exercise on muscle function, endurance, pain level, physical activity, and health related quality of life in patients with osteoarthritis of the hip.

The effects of exercise on muscle mass and the mechanisms behind the osteoarthritis, i.e., disease activity, inflammation, and cartilage degradation, are investigated in a subgroup (n=45) of the participants.

Study hypotheses: Strength training will have a greater effect on physical function and muscle strength than Nordic Walking and home based exercise; 2) Nordic Walking will have a greater effect on endurance than strength training and unsupervised home based exercise; 3) Strength training and Nordic Walking will have a greater effect on pain level and health related quality of life than unsupervised home based exercise.

ELIGIBILITY:
Inclusion Criteria:

1)Home-dwelling 60+ year old persons with primary, symptomatic hip OA who meet the clinical criteria of hip OA according to American College of Rheumatology (ACR), and who are not on a waiting list for hip joint replacement.

Exclusion Criteria:

1. symptomatic OA in the knee or the big toe,
2. joint replacement of the knee or the hip,
3. other types of arthritis, e.g., rheumatoid arthritis,
4. previous hip fracture,
5. limitation in physical function to the extent that using public transportation is impossible,
6. co-morbidity that prevents exercising,
7. physiotherapy related to hip problems within the last 3 months,
8. steroid injections in the hip joint within the last 3 months,
9. performing exercise/sports 2+ times weekly, and
10. inability to cooperate.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2009-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 2, 4 and 12 months in number of chair stands in 30 sec at 2, 4 and 12 months | Baseline, 2, 4 and 12 months

SECONDARY OUTCOMES:
Change from Baseline to 2, 4 and 12 months in isometric muscle strength (N) of the thigh and hip muscles at 2, 4 and 12 months | Baseline, 2, 4, and 12 months
Change from Baseline to 2, 4 and 12 months in lower limb extensor muscle power (Watt/kg BW) at 2, 4 and 12 months | Baseline, 2, 4, and 12 months
Change from Baseline to 2, 4 and 12 months in 6 minute walking distance (m), stair climbing time (s), 15 s marching on the spot (number of knee lifts), Timed-Up-and-Go (s) at 2, 4 and 12 months | Baseline, 2, 4, and 12 months
Change from Baseline in self-reported pain level at 2, 4 and 12 months | Baseline, 2, 4, and 12 months
  HOOS (Hip dysfunction and Osteoarthritis Outcome Score) and VAS (Visual Analogue scale)
Change from Baseline in self-reported physical activity at 2, 4 and 12 months | Baseline, 2, 4, and 12 months
  PASE (Physical Activity Scale for the Elderly) and a question from Copenhagen City Heart Study
Change from Baseline in health related quality of life at 2, 4 and 12 months | Baseline, 2, 4, and 12 months
  SF-36
Change from Baseline to 4 months in the anatomical cross sectional area (cm2) of the quadriceps femoris muscle measured with MRI. The measurements are performed in a subgroup (15 participants from each group) | Baseline and 4 months
  MRI (magnetic resonance imaging)- The anatomical cross sectional area is measured at mid-thigh level, i.e. 20 cm proximal to the tibia plateau.
Change from Baseline to 4 months in biomarkers of disease activity, inflammation, and cartilage degradation, in a subgroup (15 participants from each group) | Baseline and 4 months
  Blood samples: COMP (cartilage oligomeric matrix protein) and CRP (C-reactive protein)and Urine sample: CTX II (C-terminal telopeptide of collagen II)
Change in task specific self-efficacy from baseline to 2, 4 and 12 months | Baseline, 2, 4 and 12 months
  Self-efficacy in relation to stair climbing performance.
Change in patient global assessment from baseline to 2, 4 and 12 months. | Baseline to 2, 4 and 12 months

OTHER OUTCOMES:
Change in illness perception from baseline to 12 months | Baseline and 12 months
  Brief Illness Perception Questionnaire
Change in arthritis-specific self-efficacy from baseline to 4 and 12 months | Baseline, 4 and 12 months
  Arthritis-specific Self-efficacy Scale
Change in perceived competence from baseline to 4 and 12 months | Baseline, 4 and 12 months
  Perceived Competence Scale

CONTACTS AND LOCATIONS:
Overall Officials: Nina Beyer, Ph.D., Principal Investigator — Institute of Sports Medicine - Copenhagen & Musculoskeletal Rehabilitation Research Unit, Bispebjerg Hospital
Locations (1):
- Institute of Sports Medicine - Copenhagen & Musculoskeletal Rehabilitation Research Unit, Bispebjerg Hospital, Copenhagen, Denmark